CLINICAL TRIAL: NCT07395843
Title: Full Free-Breathing Cardiac Magnetic Resonance Imaging: Clinical Feasibility, Efficiency, and Diagnostic Concordance
Brief Title: Clinical Feasibility of Full Free-Breathing Cardiac Magnetic Resonance Imaging
Status: Completed | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Minjie Lu, Department Director, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: FB-CMR
Record Dates: First submitted 2025-12-27; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-12

CONDITIONS: FAST Scan
Keywords: free-breathing; CMR; compressed sensing; motion correction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- cine validation: compare free-breathing and breath-holding cine sequences
  Interventions: Diagnostic Test: Free-breathing CMR
- T1 mapping and LGE validation: compare free-breathing and breath-holding T1 mapping and LGE sequences
  Interventions: Diagnostic Test: Free-breathing CMR
- head-to-head validation: head-to-head comparisons of all sequences between two acquisitions
  Interventions: Diagnostic Test: Free-breathing CMR
- full free-breathing CMR: pure full free-breathing cohort

INTERVENTIONS:
Diagnostic Test: Free-breathing CMR — scan patients under free-breathing status
  Groups: T1 mapping and LGE validation; cine validation; head-to-head validation

SUMMARY:
To evaluate the feasibility, efficiency, and diagnostic concordance of a full comprehensive free-breathing cardiac magnetic resonance protocol with motion correction and sensing.

DETAILED DESCRIPTION:
This study aims to establish a large-scale, clinically oriented full free-breathing cardiac MRI framework to eliminate dependence on patient breath-holding, substantially shorten scan time, and improve patient comfort. Building on prior successful implementation of compressed sensing and motion correction techniques, the invesitgators will collaborate with the MRI vendor and sequence scientists to develop a comprehensive set of free-breathing sequences, including cine imaging, T1/T2 mapping, flow, perfusion, and late gadolinium enhancement (LGE). The study will then prospectively enroll a large, disease-diverse cohort of cardiovascular patients at Fuwai Hospital and systematically compare the full free-breathing protocol with conventional breath-hold protocols in terms of acquisition time, image quality, and agreement of quantitative parameters, thereby providing a comprehensive assessment of technical feasibility and clinical value.

ELIGIBILITY:
Inclusion Criteria:

* consecutive enrollment of patients referred for clinically indicated contrast-enhanced CMR

Exclusion Criteria:

* patients with CMR contraindications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: any patients with various cardiac diseases referred for clinically indicated contrast-enhanced CMR
Sampling Method: Non-Probability Sample
Enrollment: 605 (Actual)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
scan time | Measurements are performed within 7 days after the completion of the CMR scan.
  total CMR examination time from the scanning time of first image to the last image

SECONDARY OUTCOMES:
image quality | Measurements are performed within 7 days after the completion of the CMR scan.
  5-point Likert scale will be applied to assess image quality between two scanning methods, with a score of ≥3 considered clinically acceptable. Image quality was assessed visually using a 5-point Likert scale, defined as follows: 5 = excellent image quality; 4 = good quality with mild motion artifacts or distortion; 3 = presence of motion artifacts or distortion but sufficient image quality; 2 = fair quality with significant motion artifacts or distortion, limiting diagnostic utility; and 1 = non-diagnostic quality.
consistence of left ventricular ejection fraction | Measurements are performed within 7 days after the completion of the CMR scan.
  Linear regression and Bland-Altman analyses will be used to assess the correlation and agreement of left ventricular ejection fraction (%) from different techniques.
consistence of native T1 values | Measurements are performed within 7 days after the completion of the CMR scan.
  Linear regression and Bland-Altman analyses will be used to assess the correlation and agreement of native T1 values (ms) from different techniques.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided